CLINICAL TRIAL: NCT06526364
Title: Clinnova-MS: a Prospective Cohort Study of Patients With Multiple Sclerosis: A Trans-Regional Digital Health Effort Unlocking the Potential of Artificial Intelligence and Data Science in Health Care (Switzerland)
Brief Title: Clinnova-MS: A Prospective Cohort Study of Patients With Multiple Sclerosis (Switzerland)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Luxembourg Institute of Health (Other Government); Research Center for Clinical Neuroimmunology and Neuroscience Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01640; ko23Granziera
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
Keywords: Immune-meditated Diseases; Artificial Intelligence; Personalized medicine; Treatment change; Phenotyping; Clinnova
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (50 ml per visit), Optional: Cerebrospinal fluid (at diagnosis), stool, saliva, and hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients: MS patients, recruited from the SMSC, are annually (optional 6-monthly) assessed and additionally, perform digital measurements with the Healios+Me app continuously after baseline up to 5 years as an optional follow-up study extension.
  Interventions: Other: All participants will be asked to provide data and samples for collection and analysis.

INTERVENTIONS:
Other: All participants will be asked to provide data and samples for collection and analysis. — During the first year, data related to demographics, lifestyle, clinical examinations will be collected at baseline, at 6 months (optional) and at 12 months. PROs, cognitive and motor assessments will be performed using the Healios+Me smartphone app. Additionally, participants will be asked to provide biological samples (i.e., blood, cerebrospinal fluid and stool, saliva and hair) and imaging data (if performed as per standard of care). One unscheduled visit may be performed in case the participant comes to the hospital with the occurrence of flare or for a treatment change.
  A long-term follow-up (FU, starting from month 12 and up to 4 years after month 12) is foreseen in this study. During the long-term FU medical data are collected either every 6 month or on a yearly basis, and PROs are collected every 6 months. Whether study visits are conducted in 6- or 12-monthly intervals depends on the schedule of the study visits for the Swiss MS cohort (SMSC).

SUMMARY:
This prospective cohort study is part of the Clinnova programme and aims to (i) identify clinical imaging and omics characteristics associated with early Multiple Sclerosis (MS) and with transitioning phases to progressive MS, as well as (ii) to investigate digital biomarkers allowing the continuous clinical monitoring of those patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic disease of the central nervous system that causes a range of neurological symptoms, such as cognitive issues, fatigue, vision problems, and muscle weakness. There are two main forms: relapsing-remitting MS (RRMS) with episodes of symptoms that improve on their own, and primary progressive MS (PPMS) with chronically worsening symptoms. Many RRMS patients eventually develop secondary progressive MS (SPMS), where disability worsens without remissions. What causes MS remains unknown, but it is thought to involve genetic and environmental factors. Diagnosis and monitoring typically involve patient history, neurologic examination in combination with magnetic resonance imaging (MRI), and other tests, but these methods are costly and time-consuming. Efforts are made to develop digital tools for continuous patients monitoring.

This study is part of the Clinnova programme, aiming to collect standardized and high-quality digital health data. Clinnova-MS is a prospective cohort study including patients with early MS or those transitioning to progressive MS. Up to 100 patients, recruited from the ongoing Swiss MS cohort study, are enrolled in Basel, Switzerland. An equivalent number of patients are enrolled in other Clinnova centers, reaching at least 800 patients in total. The study aims to provide a structured and standardized highly granular dataset, allowing for the phenotyping of patients with similar patterns and disease courses. It also facilitates transnational data linkage the analysis of complex and heterogeneous data from MS patients.

The primary objective of the study is to derive a set of biomarkers that will better characterize the clinical phenotype and progression of the disease, as well as the functional impairment of MS patients at different stages. These biomarkers will aid clinicians in making informed treatment decisions for patients with early MS or those transitioning to progressive MS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Participants are willing and able to comply with the protocol, including undergoing data and samples collection as well as study visits and examinations.
* Signed informed consent form
* In possession of a Healios+Me app compatible smartphone (iOS/Android)
* Corrected close visual acuity of ≥0.5
* Hand motor skills sufficient for using a smartphone
* Ability to follow the study procedures
* Diagnosed with MS according to the revised McDonald criteria 2017, all clinical forms inclusive (clinically isolated syndrome, RRMS, SPMS, PPMS) AND early disease stages (< 3 years) OR transitioning phase to progressive disease as evaluated based on Expanded Disability Status Scale (EDSS).
* Enrolled in the SMSC at University Hospital Basel

There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS are be recruited from the ongoing clinical cohort (SMSC), where participants have annual (optional 6-monthly) visits with a well-defined assessment schedule.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Set of biomarkers | 2029
  To identify clinical, imaging and omics characteristics associated with early MS and with transitioning phases to progressive MS, a set of biomarkers is derived that allows in the future to better characterize the disease clinical phenotype and progression, the functional impairment of MS patients in different disease stages, and either associated with early MS or with transitioning phase to progressive MS, as an aid to assist clinicians in applying treatment change.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Expanded Disability Status Scale (EDSS) is assessed. The EDSS is a standardized method used to quantify disability in MS patients. The scale ranges from 0 to 10, with lower scores indicating minimal or no disability and higher scores indicating severe disability. Scores are determined based on assessments of motor function, sensory function, coordination, and other neurological functions.
9-Hole Peg Test (9-HPT) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the 9-Hole Peg Test (9-HPT) is performed. The 9-HPT evaluates manual dexterity by measuring the time it takes for the participant to move nine pegs from a box into nine holes on a board and back. Lower times indicate better dexterity and hand function, while higher times suggest greater impairment. The test will be carried out twice per hand, starting with the dominant hand, and the best performance will be used.
Timed 25-Foot Walk (T25FW) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Timed 25-Foot Walk (T25FW) is performed. The T25FW measures the time it takes for the patient to walk a distance of 25 ft (7,62 m) in their usual manner. Shorter times indicate better walking ability and mobility, while longer times suggest greater impairment.
Stroop Test (Victoria Version) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Stroop Test (Victoria Version) is performed. The Stroop Test measures processing speed and inhibition ability. First round: Participant is presented with 24 coloured dots and is asked to name the colour of the dots as fast as possible. Second round: Participant sees coloured random words (when, and, hard, over) and is asked to name the colour of each word as fast as possible. Third round: Participants is presented with 24 coloured words spelling colours (and the printed colour of the word is not the same as spelled colour), and is asked to name the printed colour as fast as possible. The test gives three scores based on the number of completed items in each round, and interference scores can be calculated.
Symbol Digit Modalities Test (SDMT) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Symbol Digit Modalities Test (SDMT) is performed. The SDMT measures information processing speed. The participant is presented with a key, matching symbols to numbers (1-9). The participant must then use this key to orally (or in written form) match symbols to digits from list during 90 seconds and the number of correctly matched symbols are counted. Higher scores indicate better cognitive processing speed and efficiency, while lower scores suggest slower processing speed and potential cognitive impairment.
Trail Making Test A&B (TMT A&B) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Trail Making Test A&B (TMT A&B) is performed. The TMT A&B evaluates information processing speed and mental flexibility. In part A, the participants are asked to connect numbers in ascending order (randomly spread out on a sheet) with a pencil as fast as they can. In part B there is an additional sequence (alphabet), also randomly spread out on the sheet. The participants must now connect switching from number to letter (e.g., 1-A-2-B-3-C…) as fast as they can. In each part, the result is measured as time to completion of the task. Lower completion times indicate better cognitive functioning, while higher times may suggest difficulties with cognitive flexibility and processing speed.
Multiple Sclerosis Inventory of Cognition (MUSIC) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Multiple Sclerosis Inventory of Cognition (MUSIC) is performed. The MUSIC evaluates various cognitive domains such as memory, attention, processing speed, and executive function. The number of correctly associated words within 1 min is measured, not counting in repetitions or missed alternations. Higher scores indicate better cognitive performance, while lower scores suggest cognitive impairment.
Digit span backwards (DSB) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Digit span backwards (DSB) is performed. The DSB assesses working memory. The tester reads out a series of random digits, which the participants must repeat starting from the last digit going to the first e.g.: tester: "1, 2, 3", participant: "3, 2, 1". The test starts with 3 digits, after each successful round (2 series of digits) the series increases 1 digit. The test goes on until the participant fails twice to reproduce the series backwards.
Rey-Osterrieth Complex Figure Test (ROCF) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Rey-Osterrieth Complex Figure Test (ROCF) is performed. The ROCF tests visuo-constructive abilities, visual memory and executive functioning (mainly planning). Participants are asked to copy and memorise a complex figure, then draw from memory after ~ 3 minutes and draw once more after ~ 30 minutes. The test proposed by Taylor (1959), which is an adapted version of the original, is used. Scoring is determined by the number of correctly drawn sub-sections of the complex figure and their position. The maximum score is 36 (18 subsections with 2 possible points per subsection (1 for correctly drawn, 1 for correctly placed). Higher scores indicate better visuospatial and memory performance, while lower scores suggest impairments in these cognitive functions.
Verbal Learn and Memory Test (VLMT) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Verbal Learn und Memory Test (VLMT) is performed. The VLMT assesses verbal learning and memory by having participants memorize and recall 15 words read aloud by a rater. This process is repeated five times with new word lists introduced between trials. The participant recalls the initial list immediately and again after a 20-30 minute delay. Scores range from 0 to 75 for learning trials and 0 to 15 for immediate and delayed recall, where higher scores indicate better memory performance and lower scores indicate cognitive challenges. The VLMT is the German precursor to the California auditory-verbal learning test.
Near vision acuity test | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Near vision acuity test is performed. The Near Vision Acuity Test measures how well a person can see and read at close distances, using a common near vision chart according to manufacturer instructions. Common charts yield ratio values from 0.1 to 1.2. The test is non-verbal. Higher scores indicate better near vision acuity, while lower scores suggest difficulties with seeing close-up details.
Contrast vision test (Pelli-Robson low-contrast chart) | Baseline and once a year for up to 5 years
  To determine the individual disease activity scores and their evolution since baseline (improvement/worsening), the Contrast vision test (Pelli-Robson low-contrast chart) is performed. This is a contrast discrimination test to detect visual disturbances (with equally large letters of decreasing contrast, organized in triplets, to be read at a distance of 1 m). The participant is asked to name the letters and the test continues until two or more errors are made for a triplet of letters. Contrast sensitivity is determined by the last triplet in which the participant can correctly name two of three letters, and the chart's log sensitivity range is from 0 to 2.25.
Short-form Food Frequency Questionnaire (SFFFQ) | Baseline and once a year for up to 5 years
  The Short-form Food Frequency Questionnaire is used to ask five questions about the typical weekly diet.
Fatigue Severity Scale (FSS) | Baseline every 6 months for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the Fatigue Severity Scale (FSS) is distributed through the Healios+Me app. The FSS is a self-report questionnaire that measures the severity of fatigue and how it has interfered with certain activities during the past 14 days. Scores range from 1 to 7 for each statement, with higher scores indicating greater severity of fatigue symptoms. Lower scores suggest milder fatigue symptoms or less impact on daily life.
Multiple Sclerosis Impact Scale (MSIS-29) | Baseline every 6 months for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the Multiple Sclerosis Impact Scale (MSIS-29) is distributed through the Healios+Me app. The MSIS-29 is a self-report questionnaire that measures the physical and psychological impact of MS during the past 2 weeks. Scores range from 0 to 100 for each subscale, with higher scores indicating a greater impact of MS on physical and psychological well-being. Lower scores suggest less impact and better quality of life in these domains.
MS Symptom Tracker | Baseline every 6 months for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the MS Symptom Tracker is integrated in the Healios+Me app. The MS Symptom Tracker consists of questions regarding symptoms experienced during the past 2 weeks.
Relapse reporting | Baseline every 6 months for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), Relapse reporting is integrated through the Healios+Me app. It allows patients to report in the app when a relapse has occurred, following a structured questionnaire.
Multiple Sclerosis Quality of Life-54 (MSQoL-54) | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the Multiple Sclerosis Quality of Life-54 (MSQoL-54) is performed. The MSQoL-54 is a self-report questionnaire on quality of life with 36 generic and 18 MS-specific items. Scores are calculated for each domain and range from 0 to 100, with higher scores indicating better quality of life. Lower scores indicate poorer quality of life in the respective domains assessed by the questionnaire.
Hospital Anxiety and Depression Scale (HADS) | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the Hospital Anxiety and Depression Scale (HADS) is performed. The HADS is a self-report questionnaire on anxiety and depression symptoms with 14 items. Each item is scored on a scale from 0 to 3, with higher scores indicating higher levels of anxiety or depression. Total scores for each subscale (anxiety and depression) range from 0 to 21, where higher scores indicate more severe symptoms of anxiety or depression.
Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 8a | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 8a is used. It consists of 8 items that ask respondents to rate their level of confidence in managing various symptoms on a scale from 1 (not at all confident) to 5 (totally confident). Higher scores indicate greater self-efficacy in managing symptoms associated with chronic conditions.
PROMIS Numeric Rating Scale v1.0 - Pain Intensity 1a | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the PROMIS Numeric Rating Scale v1.0 - Pain Intensity 1a is used. It consists of a single item where respondents rate their pain intensity on a numeric scale from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate higher levels of pain intensity reported by the individual.
PROMIS Short Form v1.1 - Pain Interference 4a | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the PROMIS Short Form v1.1 - Pain Interference 4a is used. It consists of four items that ask about the impact of pain on activities, mood, relationships, and enjoyment of life. Responses are scored on a 5-point scale ranging from 1 (not at all) to 5 (very much). Higher scores indicate greater pain interference, reflecting more significant impacts of pain on daily activities and quality of life.
PROMIS Short Form v2.0 - Cognitive Function - Abilities 8a | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the PROMIS Short Form v2.0 - Cognitive Function - Abilities 8a is used. It consists of eight items that ask about various cognitive functions such as memory, concentration, and problem-solving abilities. Responses are scored on a 5-point scale ranging from 1 (not at all) to 5 (very much). Higher scores indicate better perceived cognitive abilities, reflecting higher levels of cognitive function and capability in daily activities.
PROMIS Scale v1.2 - Global Health | Baseline and once a year for up to 5 years
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the PROMIS Scale v1.2 - Global Health is used. It includes 10 items covering physical, mental, and social health domains. Responses are rated on a 5-point scale ranging from 1 (poor) to 5 (excellent). Higher scores indicate better perceived global health, encompassing physical, mental, and social aspects of well-being.
electronic Health Literacy Scale (eHEALS) | Baseline
  To assess the quality of life and disease activity and their evolution since baseline (improvement/worsening), the electronic Health (eHealth) Literacy Scale (eHEALS) is evaluated. The eHEALS is a self-report questionnaire with 8 items measuring patients' knowledge, comfort, and perceived ability to find, evaluate, and apply electronic health information to one's health problems. It consists of 8 items rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher levels of perceived eHealth literacy, reflecting greater confidence and ability in using online health information effectively.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Granziera, Prof., Principal Investigator — Research Center for Clinical Neuroimmunology and Neuroscience Basel (RC2NB)
Locations (1):
- Research Center for Clinical Neuroimmunology and Neuroscience Basel (RC2NB), Basel, Switzerland

REFERENCES:
- See also: CLINNOVA website — https://www.clinnova.eu/en/